CLINICAL TRIAL: NCT04795297
Title: Observational Study of Basal Cell Carcinoma Operated at Montpellier University Hospital and Millau Hospital From February 2020 to February 2021 - Study of Correlation Between Localisation and Recurrence, and Other Criterias
Brief Title: Observational Study of Correlation Between Recurrent Basal Cell Carcinoma and Localisation
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0156
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Basal Cell Carcinoma
Keywords: Resection of BCC (Basal Cell Carcinoma); Recurrence of BCC (Basal Cell Carcinoma); Localisation
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent BCC: recurrent BCC
- resected BCC: resected BCC

SUMMARY:
.During one year all the resected basal cell carcinomas (BCC) analyzed in Montpellier University Hospital Anatomopathology unit were included in this study. Localisation and histological characteristics were collected. All the recurrences of BCC were searched from the medical records (or histopathology request form).

From 804 BCC, 48 were recurrent BCC with or without complete first resection. Patients with recurrent BCC were contacted to obtain agreement and more informations about the first resection and some clinical informations like sun exposure and phototype.

The statistical analysis focused on the localisation of recurrent BCC (with a complete first resection) compared to localisations of primary BCC in this population. The goal was to identified localisations with an increased risk of recurrences.

ELIGIBILITY:
Cohort :

Inclusion criteria:

- Patients with resected BCC

Exclusion criteria:

* Biopsies of BCC,
* revised surgery of incomplete resection.

Cases :

Inclusion criteria:

-Recurrent BCC with complete first resection

Exclusion criteria:

- Recurrent BCC with incomplete first resection, Patients with Gorlin syndrome (a genetic disease that increase risk of BCC)

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort :
  All the resected BCC during one year in Montpellier University Hospital and Millau Hospital (both analyzed in anatomopathology unit in Montpellier University Hospital).
  Cases :
  All the cases of recurrent BCC, found after research in medical records or histopathology request form.
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
- Determined For each localisation the number of primary and recurrent BCC and analysis of localisation with higher risk of BCC | 1 day
  - Determined For each localisation the number of primary and recurrent BCC and analysis of localisation with higher risk of BCC

SECONDARY OUTCOMES:
Analysis of correlation between localisation and histology characteristics | 1 day
  Analysis of correlation between localisation and histology characteristics
Analysis of correlation between histological type and recurrence risk | 1 day
  Analysis of correlation between histological type and recurrence risk
Analysis if there is a difference between first resection histological type and the recurrent histological type | 1 day
  Analysis if there is a difference between first resection histological type and the recurrent histological type

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Pons, Resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC